CLINICAL TRIAL: NCT05643924
Title: The Use of the COM-B Questionnaire to Determine the Psychological and Behavioural Barriers to Adherence in Patients with Asthma
Brief Title: COM-B Asthma Questionnaire
Acronym: COM-B
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: University of Portsmouth (Other)
Responsible Party: Sponsor
Other Study IDs: 300735
Record Dates: First submitted 2022-11-21; First posted 2022-12-09 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Asthma
Keywords: Asthma; Adherence; Behaviour and psychological barriers; COM-B; Inhaler; Theoretical Domains Framework; Behaviour change
MeSH Terms: conditions — Asthma; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients diagnosed with Asthma

SUMMARY:
Asthma is a common lung condition that cannot be cured, although usually it can be effectively controlled with available treatments. Yet, it is well recognised that 70% of patients are non-adherent to their asthma treatment.

Personalising treatment by offering the most relevant interventions based on the patient's psychological/behavioural needs results in great success. However, health care providers have limited available resources to deliver a patient-centred approach to their psychological/behavioural needs, resulting in a current one-size-fits-all strategy due to the non-feasible nature of existing surveys.

The solution would be to provide health care professionals with a clinically feasible questionnaire that identifies the patients personal psychological/behavioural factors to adherence.

DETAILED DESCRIPTION:
Asthma is a common lung condition affecting over 5.4 million people in the UK, for some people, it can affect daily activities and lead to life-threatening consequences. (Asthma UK 2020). Asthma cannot be cured, but it can usually be effectively controlled with available treatments provided they are taken as recommended; however, it is well recognised that up to 70% of patients do not take their asthma treatments as recommended (are non-adherent). This is perhaps not unexpected in the context of a chronic condition requiring daily treatments, which must be taken even when the person feels well. People may also have concerns about using long-term medicines (including steroid inhalers,) or there may be other psychological/behavioural barriers to adherence. Non-adherence to asthma treatments results in poor asthma control with persisting asthma symptoms, more frequent asthma attacks and greater impairment in quality of life. There are also significant economic implications associated with 'wasted' medications and additional healthcare utilisation, such as doctors' appointments and visits to A&E, which contribute to the overall cost of asthma care in the UK, exceeding £1 billion per year.

Health care professionals play an important role in engaging and educating patients about the importance of their asthma treatments, monitoring asthma control and identifying whether a patient is adherent or not. Adherence is complex involving (1) being able to start prescribed medications; (2) taking the medications as prescribed (correct dose, inhalation technique, and frequency); and (3) persistence (obtaining refills to maintain adherence over time). There are limited resources available in a busy health care setting to ensure a complete understanding of each individual's psychological/behavioural barriers, with a one-size-fits-all approach adopted with limited success. As such, there is a persistent unmet need for a tool that can effectively identify these barriers to adherence in a clinical setting, allowing health care professionals to provide effective personalised treatments for non-adherence in patients with asthma.

It is important that the psychological needs of patients can be easily assessed to allow for the patients' personal needs to be understood, promoted, improved, and supported (Lyons & Chamberlain, 2006). When focusing on adherence behaviour, currently, the tools available are questionnaires, but these are long and complex to complete. The COM-B model is a new questionnaire that is shorter and easier for patients to complete. It involves three key components: Capability, Opportunity, and Motivation (Michie et al., 2017). These components were grouped from current health psychological theories of behaviour and behaviour change, therefore, providing a theoretical lens through which to view the physical capability, psychological capability, physical opportunity, social opportunity, reflective motivation, and automatic motivation of individuals. The information gathered from the COM-B framework can then be used to identify what needs to change for a behavioural change intervention to be successful (Michie, Van Stralen & West, 2011).

An easily accessible theory-based tool (a questionnaire) that can identify the psychological and behavioural barriers of patients with asthma who are non-adherent with their treatment is urgently required. This will allow healthcare professionals to use effective personalised interventions to support improved medication use whilst recognising and meeting the psychological needs of patients with asthma. Additionally, the Covid pandemic has changed the way people with asthma access their care with a move to remote consultations and questionnaire completion. The COM-B questionnaire may well be suitable for this approach. Still, it is essential to assess digital readiness in this population to understand whether this is feasible and inform the design of future studies if the COM-B questionnaire proves to be successful.

Primary Objective:

- To assess the short COM-B questionnaire's capacity to detect patients' perceived psychological and behavioural barriers to adherence in asthma patients.

Secondary objectives:

* To determine whether the COM-B questionnaire can be employed in a busy clinical setting.
* To explore the key psychological and behavioural barriers indicated by the COM-B questionnaire and adherence to treatment in patients with confirmed asthma with heterogenous severity.

Exploratory objectives:

* To assess the relationship between a patient's capability, opportunity, motivation, and asthma phenotype, including clinical, biological, psychosocial, and behavioural components.
* To explore the associations between the COM-B questionnaire responses and digital readiness.

This study will employ a cross-sectional survey design. It will be delivered online through the REDCap platform. One hundred and forty six participants will be recruited when attending their routine clinical review with the asthma service or whilst an inpatient at Queen Alexandra Hospital - this is based on a sample size that has been calculated using GPower software. Participants will be asked to complete a set of questionnaires that takes no longer than 20 minutes to complete. The questionnaires used have all been verified, and permission to use them in the study has been given. They will assess:

1. Psychological and behavioural barriers that may affect the participant being able to take their asthma treatments as recommended: the brief COM-B questionnaire (which is being validated as part of this study) and the 61-item Theoretical Domain Framework Questionnaire (TDFQ)
2. Their asthma symptoms and how well controlled their asthma is (ACQ-6); The impact their asthma has on their quality of life (mini-AQLQ); the level of anxiety and/or depression they may be experiencing (Hospital Anxiety and Depression Scale). All of these questionnaires are used routinely at clinic reviews
3. Their use of technology at home and any challenges they face with this: digital readiness questionnaire.

Patient data that is routinely collected, such as demographics, asthma characteristics, asthma control, and medication regimen, will be recorded on an electronic data capture form (e-CRF) through the REDCap platform by a member of the research team.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Willing and able to give informed consent for participation in the study.
* Diagnosis of asthma confirmed by a healthcare professional and requiring maintenance asthma treatment, including an inhaled corticosteroid

Exclusion Criteria:

* Unable to comprehend the study and provide informed consent, e.g., insufficient command of English in the absence of someone who can adequately interpret.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All people with a diagnosis of asthma, under the care of the asthma service at Portsmouth Hospitals University NHS Trust will be invited to participate in this study. This will include recruitment from both primary and secondary care sites. In addition, both outpatients and inpatients will be approached and invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Can the COM-B questionnaire detect a patient's perceived psychological and behavioural barriers to adherence | 3 Years
  Comparisons of the (1) short COM-B questionnaire (2) 61-item Theoretical Domain Framework Questionnaire to assess content validity. A low score on the COM-B questionnaire and the Theoretical Domains Framework Questionnaire indicates that the individual is experiencing a barrier based on that source of behaviour domain.

SECONDARY OUTCOMES:
Can the COM-B questionnaire be used in a clinical asthma pathway? | 3 Years
  The total number of questionnaires distributed and the proportion of completed questionnaires compared to the 61-item Theoretical Domain Framework Questionnaire and the asthma control questionnaire (ACQ).
To explore the key psychological and behavioural barriers indicated by the COM-B questionnaire and adherence to treatment in patients with confirmed asthma with heterogenous severity | 3 Years
  Compare responses between capability, opportunity and motivation (COM-B components) with levels of adherence measured by:
  1) Medicines Possession Ratio (MPR)

OTHER OUTCOMES:
Exploring the associations between the COM-B questionnaire responses and asthma phenotype, including clinical, biological, psychosocial and behavioural components | 3 Years
  Compare responses between capability, opportunity and motivation (COM-B components) with variables including (but not limited to):
  1. Type of asthma (T2 or non-T2 defined by the presence of a T2 inflammatory signal assessed using FeNO and/or peripheral blood eosinophil count)
  2. Asthma severity using BTS/SIGN stage
  3. Level of asthma control assessed using the ACQ6 questionnaire (a score of ≥1.5 reflects poor asthma control and number of severe exacerbations in preceding 12 months
  4. Quality of life measured using the mini AQLQ score
  5. Number of co-morbidities
  6. The complexity of treatment (number of inhaled doses/day, total number of medications taken each day)
  7. Item responses from the digital readiness questionnaire
Explore the associations between the COM-B questionnaire responses and digital readiness | 3 Years
  Compare responses between capability, opportunity and motivation (COM-B components) and scores of the digital readiness scale. Low COM-B questionnaire scores indicate that interventions are needed, and low digital readiness scores indicate that the individual will struggle with digital technology.

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals University NHS Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munns A, Wiffen L, Brown T, Fasulo A, Chauhan M, D'Cruz L, Kaklamanou D, Chauhan AJ. Capability, Opportunity, and Motivation Model for Behavior Change in People With Asthma: Protocol for a Cross-Sectional Study. JMIR Res Protoc. 2023 Jul 6;12:e44710. doi: 10.2196/44710. PMID 37410518